CLINICAL TRIAL: NCT02305550
Title: A Proof of Concept Study of Electrical Discharge Produced Nitric Oxide for Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Anesthesiologist and Intensivist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: eNO for inhalation
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hypertension, Pulmonary
Keywords: Nitric Oxide
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electrical synthesis nitric oxide (Experimental): Participants will breath 20 minutes of electrical pulsed plasma discharge synthesis of nitric oxide at 25 parts per million
  Interventions: Device: electrical pulsed plasma discharge synthesis of nitric oxide

INTERVENTIONS:
Device: electrical pulsed plasma discharge synthesis of nitric oxide — An NO generator was designed and developed by electrical pulsed plasma discharge nitric oxide from atmospheric nitrogen and oxygen. This generator has been fabricated by the investigators and it is not commercially available.

SUMMARY:
Study Design: This is a two-part physiological for a device feasibility. Both studies are proof of concept descriptive pilot studies.

The FIRST PART is a study of healthy volunteers and the SECOND PART of patients with pulmonary hypertension at routine cardiac catheterization laboratory (CATH-LABORATORY).

Volunteers and patients will be enrolled sequentially; there is no group randomization.

Overall hypothesis of this device feasibility study: To test a lightweight and portable method of synthesizing therapeutic levels of inhaled nitric oxide from air by electrical pulsed discharge.

DETAILED DESCRIPTION:
Background. Inhaled nitric oxide is routinely used to treat acute pulmonary hypertension in infants, children and adults. By 2014 it has been estimate about 500,000 US patients have been treated with nitric oxide, with only the rare complication of methemoglobinemia reported at high inhaled doses.

Rationale. The investigators explored novel alternative lightweight and economical methods of local nitric oxide production. In particular the investigators synthesized nitric oxide from air by an electrical pulsed plasma discharge. After 2 years of study the investigators have designed and produced a prototype of a device synthesizing nitric oxide from air with low levels of nitrogen dioxide and ozone. After completing experimentation in lambs, the investigators now plan to study nitric oxide generators in a proof of concept clinical study.

Design of the study: The study is comprised of two parts:

1. HEALTHY volunteer study, and
2. CATH-LABORATORY study in patients.

The study will be conducted at low levels of breathing nitric oxide, 25 parts per million of nitric oxide, for 20 minutes to comply with the threshold of the Environmental Protection Agency (EPA) for daily work exposure.

The first portion of the study will be carried out in 6 healthy volunteers breathing 25 parts per million of nitric oxide. After this first part, the investigators will proceed to the second portion of the study and enroll 6 patients with pulmonary hypertension undergoing scheduled testing with a nitric oxide-pulmonary vasodilator response (CATH-LABORATORY study).

ELIGIBILITY:
FIRST PART OF THE STUDY: HEALTHY VOLUNTEER STUDY (n=6 volunteers)

Inclusion Criteria:

* Have a government photo identity card;
* Age < 40 years old;
* Body mass index (BMI) <28 kg/m2 and >18 kg/m2;
* Feel well the day of nitric oxide testing;
* Normal physical exam

Exclusion Criteria:

* Psychiatric disturbances such as anxiety, depression, schizophrenia requiring pharmacological treatment or hospitalization in the last year;
* Systemic disease with or without any functional limitation; including controlled hypertension and controlled diabetes without systemic effects;
* Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin, or less than six weeks postpartum;
* Active smoking, volunteers may be enrolled if they quit smoking for more than 1 year;
* Excess alcohol use: more than ½ L/day of wine consumption or equivalent;
* Any current use of a medication other than: Over-the-counter oral medications, herbal remedies, nutritional supplements, and oral contraceptives;
* Currently enrolled in another research study.

SECOND PART OF THE STUDY: CATH-LABORATORY STUDY (n=6 cath laboratory subjects)

Inclusion criteria:

* Have a government photo identity card;
* Diagnosis of Pulmonary Arterial Hypertension, Group I, III, IV and V, as defined by the National Heart Lung and Blood Institute classification.
* Known positive responder to inhaled nitric oxide
* Wedge pressure ≤15 mmHg at baseline
* Pulmonary arterial pressure (mean) greater than or equal to 40 mmHg
* Scheduled Cath Lab testing for right heart catheterization to assess pulmonary vasodilator capacity

Exclusion Criteria:

* Psychiatric disturbances such as anxiety, depression, schizophrenia requiring pharmacological treatment or hospitalization in the last year;
* Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin, or less than six weeks postpartum;
* Left ventricular failure for which breathing nitric oxide is contraindicated;
* Patients with diagnosis of congenital or acquired methemoglobinemia reductase deficiency;
* Currently enrolled in another research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 20 minutes
  Percent change in oxygen saturation (HbO2/totHb)
Methemoglobin | 20 minutes
  Percent change in methemoglobin levels (metHb/totHb)
Carboxyhemoglobin | 20 minutes
  Percent change in carboxyhemoglobin levels (COHb/totHb)

SECONDARY OUTCOMES:
Pulmonary artery pressure | 20 minutes
  Change in pulmonary artery pressure (mmHg)
Cyclic guanosine monophosphate | 20 minutes
  Percent change in plasma cyclic guanosine monophosphate (measured over baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Malhotra R, Hess D, Lewis GD, Bloch KD, Waxman AB, Semigran MJ. Vasoreactivity to inhaled nitric oxide with oxygen predicts long-term survival in pulmonary arterial hypertension. Pulm Circ. 2011 Apr;1(2):250-258. doi: 10.4103/2045-8932.83449. PMID 22020367
- [Background] Frostell C, Fratacci MD, Wain JC, Jones R, Zapol WM. Inhaled nitric oxide. A selective pulmonary vasodilator reversing hypoxic pulmonary vasoconstriction. Circulation. 1991 Jun;83(6):2038-47. doi: 10.1161/01.cir.83.6.2038. PMID 2040056